CLINICAL TRIAL: NCT05964764
Title: A Pragmatic, Prospective, Multicentre Study for the Validation of the Scandinavian Guidelines for Minor and Moderate Head Trauma in Children
Brief Title: Validation of the Scandinavian Guidelines for Minor and Moderate Head Trauma in Children
Acronym: SHIPP
Status: Recruiting | Type: Observational
Sponsor: Halmstad County Hospital (Other)
Responsible Party: Principal Investigator, Fredrik Wickbom, Principal Investigator, Halmstad County Hospital
Other Study IDs: 220871
Record Dates: First submitted 2023-06-22; First posted 2023-07-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples Without DNA — In a subgroup of patients (target n=1000) a blood and saliva sample for postponed analysis of biomarkers in TBI will be obtained after written informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Head injuries are common among children and adolescents, with many of them assessed in emergency departments each year. Most children recover fast, with full resolution of symptoms as headache, dizziness or fatigue. A few, however, develop life-threatening complications (such as bleedings in/around the brain). It can be difficult to swiftly and accurately identify these patients in the emergency department. To aid in this task, decision support tools has been developed.

The goal of this observational study is to evaluate a Scandinavian tool developed to aid in management of children with head injuries seeking care in an emergency department.

The main research question is:

- Are the Scandinavian guidelines for management of mild and moderate head trauma in children sensitive for patient-important outcomes?

Patients will be given the same treatment and recommendations for their head injury no matter if they participate or not in the study, as there is no intervention/ treatment group.

The doctor or nurse managing the child will collect information on patient history, signs and symptoms in the emergency department and management in an electronic case report form. Information on how the recovery period is collected both from medical records >1 month after the emergency department visit, as well as via electronic questionnaires sent to the guardian at 1 month, 3 months and 4 months after the injury via e-mail and/or text message. Long-term outcome will also be examined (>6 months).

DETAILED DESCRIPTION:
Design:

This is a pragmatic, prospective, multicentre, observational study of children presenting with mild or moderate traumatic brain injury (TBI) in a general or paediatric emergency department (ED) at hospitals in Scandinavia. A complete data set for analysis including predictor variables and outcome data for the six guidelines included in the study will be registered (SNC2016, PECARN, CATCH, CHALICE, PREDICT, NICE23). There are no interventions as the study is observational. Attending physicians and nurses are instructed to manage children in accordance with the hospital's ordinary guidelines and follow local treatment traditions.

Study setting and population:

The study will be set in Sweden and Norway. Hospitals with different trauma capacities will participate; invitations are sent to units which on daily basis mange children with TBI in their department. Efforts are made to establish a representative distribution in participating centres. The coordinating centre is Halmstad Hospital in southern Sweden.

Data registration and follow-up:

Information on management in the emergency department including patient characteristics, injury type and mechanism, patient history, clinical examination results and current medications will be prospectively documented in a web- based case-report form by the triage nurse and/or physician on call.

One month after trauma, the local study coordinator will assess medical records and journals, screening for outcome measures as well as CT findings, when applicable. A follow-up questionnaire will be sent to guardian(s) 1 month, 3 months and 4 months after the child ́s head injury via e-mail and/or text message (long-term follow up at >6 months). Reminders will be re-sent if no answer is received, primarily by e-mail and then twice by text message.

All data will be registered in via web-based case report forms in Entermedic (Entergate AB). Pseudo-anonymized data will be extracted from database and imported to IBM SPSS® Statistics software version 28 for statistical analysis.

Biomarkers:

A sub-study on patients with intermediate risk for intracranial injury and GCS 14-15, in selected study centres will explore biomarkers as predictors for intracranial injury. Venous blood, capillary blood and saliva sample is sampled from the patient in the ED after written informed consent. Sampling is done within 12 hours from the time of the injury. Analysis of biomarker S100B and others, not yet specified, will be analysed in batch at end of sub-study period.

CT examinations:

CT scans are analysed by a board-certified radiologist on the centre where the exam is performed.

Statistics:

The accuracy of the (SNC) guidelines to predict the primary endpoint will be assessed by 95% confidence intervals (CI) for sensitivity, specificity, likelihood ratio, negative predictive value (NPV) and positive predictive value (PPV). Test performance for other internationally recognized clinical decision rules (PECARN, CATCH, CHALICE, NICE, PREDICT) will also be calculated both in application cohorts (defined by each rule specific inclusion and exclusion criteria) and in comparative cohorts (minor head injury cohort = all patients with GCS 13-15; all patient cohort). When assessing CDRs other than SNC16, both rule specific endpoints and in-study defined endpoints will be tested. Secondary endpoints will be assessed using the same methods. Biomarker analysis results in ROC curves for sensitivity / specificity and from these are specific cut-offs that maximize performance for negative predictive value (i.e., to avoid unnecessary CT examinations and/or admission) derived.

Sample size:

The investigators aim to include 5,300 children, but not more than more than 4 years of active enrolment.

Ethics:

Ethical approval was granted from the Regional Ethical Review Board in Lund (approval number 2017/238) and Ethical Review Board in Norway (approval number 1085). Informed verbal consent will be obtained and registered. Patients' data and social security number will be stored and handled accordingly to European Union General Data Protection Regulation (GDPR 2016/679) and applicable Swedish laws.

A detailed protocol describing study methodology and statistical methods will be published before end of inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years.
* Minor and moderate blunt head trauma (GCS 9 - 15) seeking medical assessment in an emergency department at a study hospital in Sweden or Norway.
* Within 24 hours of trauma.
* Informed oral consent from one guardian, and child if older than 14 years old, after receiving oral and written information about study.

Exclusion Criteria:

* Patient and/or guardian does not wish to participate in the study.
* Patient included in other study that may affect the management/treatment in the emergency department.
* Penetrating head injury (as those will always receive a CT scan).
* Suspected child abuse / non-accidental trauma (NAT) denoted as suspected child abuse where the social services are informed (as they will always receive a CT scan).
* The patient is not a citizen in the participating country and hence difficult to follow up.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Target population is children in Scandinavia with recent minor and moderate head trauma seeking care on emergency departments within participating in study.
Sampling Method: Non-Probability Sample
Enrollment: 5300 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with "clinically important intracranial injury (CIII)" | Within 1 week of injury.
  Defined as a composite variable of death, neurosurgery, admission to hospital ward two (2) days or more due to head injury or intubation one (1) day or more due to pathological traumatic CT findings.

SECONDARY OUTCOMES:
Number of participants with death due to head injury | Within one week; within 3 months.
  Defined as death as consequence of the TBI
Number of participants with neurosurgery due to TBI | Within 1 week of injury.
  Defined as need for any neurosurgical procedure or intervention, including sedation and intubation with controlled ventilation for non-surgical injuries such as diffuse axonal injury.
Number of participants with CT findings | Within 1 week of injury.
  Defined as a possibly trauma-related intracranial finding on CT-scan, such as cranial fractures or acute intracranial haemorrhage.
Number of participants with significant CT findings | Within 1 week of injury.
  Defined as a possibly trauma-related intracranial finding on CT-scan, such as cranial fractures or acute intracranial haemorrhage, but not including undislocated skull fractures
Concentration of specific biomarkers in serum and saliva | Sampling at admission to the emergency department
  Biomarker concentration (S-100B, GFAP, UCH-L1, NSE, tau, NF(H and L), H-FABP, SNTF, MBP, miRNAs, IL-10, BTP, SBDP145, MMP9, HGF, IL-6, OPN, SAA, SICAM, leptin, copeptin, fibrinogen, d-dimer, ICAM, VCAM, IL-12, eotaxin, TNFR2 in a group of patients with TBI and GCS 14-15 in ED.
Number of participants admitted to in-hospital observation > 2 days | Within 3 months from injury
  Admission to a hospital ward two (2) days or more due to TBI.
Number of participants admitted to in-hospital observation | Within 3 months from injury
  Admission to a hospital ward due to TBI, irrespective of duration of observation
Number of participants with extended "clinical observation in ED" | Within the first day (24 hours) of injury
  Prolonged clinical observation in ED due to TBI
Duration of clinical observation | Within 1 week of injury.
  Duration of clinical observation (time in ED or time in ED and in-hospital ward)
Number of participants intubated due to TBI | Within 3 months from injury
  Endotracheal intubation due to TBI
Duration of intubation due to TBI | Within 3 months from injury
  Duration of intubation categorised as <6h, 6-12 h, 13-24h, 25-48 h, 49h-1 week and >1 week.
Number of participants referred for cranial CT (cCT) due to head injury. | Within 3 months from injury
  Referred for cCT due to head injury
Number of participants referred for a follow up (re-)cCT due to clinical deterioration. | Within 3 months from injury
  Referred for re-cCT due to clinical deterioration.
Number of participants referred for a cCT due to clinical deterioration during prolonged observation (in ED or on ward). | Within 3 months from injury
  Referred for (primary) cCT due to clinical deterioration during prolonged clinical observation.
Number of participants with need for sedation or intubation during cCT exam | Within 3 months from injury
  All ages and stratified 0-4 years, 5-14 years and >14 years. Sedation is defined as positive if participant has received a sedative agent (for example propofol or midazolam) during CT scan.
Number of participants with presence of outcome as defined by CATCH-rule ("need for neurological intervention" or "brain injury on CT" ) | Within one week from trauma
  Need for neurological intervention is defined as either death within 7 days secondary to the head injury or need for any of the following procedures within 7 days: craniotomy, elevation of skull fracture, monitoring of intracranial pressure, or insertion of an endotracheal tube for the management of head injury.
  Brain injury on CT defined as any acute intracranial finding revealed on CT that was attributable to acute injury, including closed depressed skull fracture.
Number of participants with presence of outcome as defined by PECARN-rule ("clinically important TBI"). | Within one week from trauma
  Clinically important TBI is defined as death from TBI, neurosurgical intervention for TBI (intracranial pressure monitoring, elevation of depressed skull fracture, ventriculostomy, haematoma evacuation, lobectomy, tissue debridement, dura repair, or other), intubation of more than 24 h for TBI or hospital admission of 2 nights or more for TBI in association with TBI on CT.
Number of participants with presence of outcome as defined by CHALICE-rule ("clinically significant intracranial injury" or "presence of skull fracture" or "admission to hospital"). | Within one week from trauma
  Clinically significant intracranial injury is "defined as death as a result of head injury, requirement for neurosurgical intervention, or marked abnormality on CT.
Number of participants with presence of outcome as defined by PREDICT-rule ("clinically important intracranial injury in need for intervention"). | Within one week from trauma
  Clinically important intracranial injury in need for intervention is defined as neurosurgery and/or intensive care due to TBI.
Number of participants with presence of outcome as defined by NICE23-rule ("clinically important traumatic brain injury") | Within one week from trauma
  Clinically important traumatic brain injury is assumed to be the same as in PECRAN, hence defined as death from TBI, neurosurgical intervention for TBI (intracranial pressure monitoring, elevation of depressed skull fracture, ventriculostomy, haematoma evacuation, lobectomy, tissue debridement, dura repair, or other), intubation of more than 24 h for TBI or hospital admission of 2 nights or more for TBI in association with TBI on CT.
Number of participants reassessed or readmitted due to TBI | Within four weeks from trauma
  Reassessed and sent home from ED, or admitted from ED after reassessment due to prior TBI.
Number of participants transported to other hospital due to TBI | Within 3 months from injury
  Transport to other hospital due to TBI, irrespective of cause or way of transportation.
Time to full recovery | <1 week, 1 week, 2 weeks, 3 weeks, 1 month, 2 months, 3 months, not recovered at 3 months
  Time to full recovery from TBI
Clinicial utility SNC16 rule | At admission to the emergency department.
  Experienced utility of the SNC16-rule when applied hypothetically on the participating child with TBI, by the managing doctor. Assessed on a 7-step Likert scale.

OTHER OUTCOMES:
Participant rating on GOS-E PEDS Score | 3 months after injury
  Clinical outcome according to GOS-E PEDS (paediatric Glasgow Outcome Scale extended version), score 1-8 (higher score indicate worse outcome), assessed by parent.
Participant rating on Post Concussion Symptom Inventory - Parent (PCSI-P) assessment | 3 months after injury.
  Clinical outcome on PCSI-P assessed by parent on a 20-item scale. Each item assessed on a 7-point scale (0 = not a problem, 6 = severe problem).
Participant rating on Mental Fatigue Scale | 1 month and 4 months after injury.
  Clinical outcome on modified Mental Fatigue Scale assessed by parent. 15 items assessed 0 - 2/3. Higher value indicates a higher degree of severity. One question on variation of symptoms over day. One question on pre-injury status.
Long-term outcome | 5 years post TBI
  Assessment of remaining post concussive symptoms at 5 years after TBI. Assessed by GOS-E PEDS, PCSI-P and Mental Fatigue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Undén, MD, PhD., Study Chair — Region Halland and Lund University, Sweden
Locations (16):
- Haukeland Universitetssjukehus, Haukeland, Norway
- Sweden (15):
  - Alingsås Lasarett, Alingsås
  - Mälarsjukhuset i Eskilsstuna, Eskilstuna
  - Drottning Silvias Barnsjukhus, Gothenburg
  - Halland Hospital Halmstad, Halmstad
  - Länssjukhuset Ryhov, Jönköping
  - Lasarettet i Ljungby, Ljungby
  - Skåne University Hospital, Lund, Lund
  - Skånes Universitetssjukhus Malmö, Malmo
  - Mora Lasarett, Mora
  - Örebro Universitetssjukhus, Örebro
  - Astrid Lindgren Childrens Hospital, Solna, Stockholm
  - Norra Älvsborgs Länssjukhus, Trollhättan
  - Norrland University Hospital, NUS, Umeå
  - Halland Hospital Varberg, Varberg
  - Ystad Lasarett, Ystad

IPD SHARING:
Plan to Share IPD: Yes
Sharing of de-identified data for all primary and secondary outcome measures will be considered on individual basis after main and secondary analysis has been completed.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available on reasonable request up to 10 years after study completion.
Access Criteria: Investigators whose proposed use of the data has been approved by the study review committee and sharing of requested data is permitted by Swedish and European law.

REFERENCES:
- [Derived] Wickbom F, Thornberg S, Sotoca Fernandez J, Silfver R, Marklund N, Unden J; Scandinavian Neurotrauma Committee. Comparison of predictive tools for management of paediatric mild TBI: a prospective cohort study. EClinicalMedicine. 2025 Sep 9;88:103484. doi: 10.1016/j.eclinm.2025.103484. eCollection 2025 Oct. PMID 40979218
- [Derived] Wickbom F, Calcagnile O, Marklund N, Unden J. Validation of the Scandinavian guidelines for minor and moderate head trauma in children: protocol for a pragmatic, prospective, observational, multicentre cohort study. BMJ Open. 2024 Apr 3;14(4):e078622. doi: 10.1136/bmjopen-2023-078622. PMID 38569695
- See also: Study information page — http://www.shipp.se/